CLINICAL TRIAL: NCT07374107
Title: MIHRA - Patient-Rooted Insights for Shaping Myositis Science (PRISMS) - A Qualitative Study of Patient-voiced Research Priorities Across Rare Myositis Diseases
Brief Title: MIHRA - Patient-Rooted Insights for Shaping Myositis Science (PRISMS)
Acronym: MIHRA-PRISMS
Status: Recruiting | Type: Observational
Sponsor: Myositis International Health & Research Collaborative Alliance Foundation (Other)
Collaborators: MIHRA Patient Advisory (Unknown); Myositis Australia (Unknown); CureJM (Unknown); The Myositis Association (Unknown); The Dutch Myositis Association (Unknown); The Swedish Myositis Association (Unknown); Myositis UK (Unknown); The German Myositis Association (Unknown); CARRA - Childhood Arthritis & Rheumatology Research Alliance (Unknown); PReS - Paediatric Rheumatology European Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: MIHRA - 001; PRISMS (Other: MIHRA Foundation)
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: IBM; IIM; Myositis; Inflammatory Myopathy; Dermatomyositis; Dermatomyositis, Juvenile; Anti-synthetase Syndrome; Immune-Mediated Necrotizing Myopathy; Polymyositis; Inclusion Body Myositis; Juvenile Myositis; Juvenile Dermatomyositis
Keywords: myositis; rare diseases; patient priorities; patient engagement; patient initiated; patient research partners; qualitative research; mixed methods research; research priorities
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis; Myositis, Inclusion Body; Rare Diseases; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals living with a myositis disease: Adults and children with a clinician diagnosis of an inflammatory myopathy (and optionally caregivers/partners) will express their priorities and insights regarding regarding research priorities across myositis diseases.
  Interventions: Other: No intervention - qualitative and mixed methods investigations

INTERVENTIONS:
Other: No intervention - qualitative and mixed methods investigations — No Intervention

SUMMARY:
Myositis diseases are each rare diseases. As in other rare diseases, people living with myositis diseases face physical and psychosocial challenges that may not be recognized in current research priorities. The PRISMS study is a global investigation that collects patient perspectives through (mostly online) methods of open-ended questions, community forums and survey to identify the most pressing research concerns as identified by patients. Findings will be analyzed to create a patient-voiced set of research priorities that can guide the direction of research and help inform funding decisions across myositis diseases.

Potential participants can express interest via https://mihrafoundation.org/mihra-programs/mihra-patient-contact-registry/

DETAILED DESCRIPTION:
This is a patient-initiated observational qualitative (largely online) study engaging people living with myositis diseases (and optionally their care partners) in mixed methods applications to elicit patient-voiced research priorities. Participants will be purposively sampled to ensure representation across myositis subtypes and key demographic/clinical characteristics.

Methods include open-ended narratives, interactive focus groups and forums, rating and ranking to establish degree of importance and priorities.

Results will include a structured set of patient-voiced priority topics/questions and a draft framework for downstream consensus processes and research agenda setting.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Have a clinician diagnosis of an idiopathic inflammatory myopathy or be a care partner or parent of a person living with an idiopathic inflammatory myopathy.
* Participants who may have signed up through the MIHRA Patient Contact Registry https://mihrafoundation.org/mihra-programs/mihra-patient-contact-registry/

Exclusion Criteria:

* Under the age of 7 years old
* Do not have a diagnosis of an inflammatory myopathy

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children living with an idiopathic inflammatory myopathy recruited through self-referral (prompted by clinic notices/ patient organization newsletters / /advocacy communities / social media / internet searches ) to provide perspectives on research priorities.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Patient-voiced research priority topics | At completion of narrative, focus group forum or survey, up to 90 minute
  Number and distribution of coded priority domains identified from data collection that has been stratified by disease type, through thematic analysis (codebook refined iteratively) with subsequent assigned degree of importance and ranked priority.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Ann Saketkoo, MD, MPH, Study Chair — MIHRA Foundation
Locations (1):
- MIHRA Foundation - This is a GLOBAL STUDY, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified aggregate themes/coded domains may be shared; raw transcripts/audio will not be shared.
Supporting Information: CSR, Analytic Code
Time Frame: Data will become available immediately and remain available
Access Criteria: Through publication and by contacting info@MIHRAfoundation.org
URL: http://MIHRAfoundation.org

REFERENCES:
- [Background] Saketkoo LA, Paik JJ, Alexanderson H, Dimachkie MM, Ernste FC, Naddaf E, Shafranski B, Gupta L, Mecoli CA, Saygin D, Albayda J, Basharat P, Day JA, Valenzuela A, Bromley R, de Groot I, Edison SE, Lanis A, Lood C, Regardt M, Yi BY, Benitez AC, Chinoy H, Christopher-Stine L, Isenberg DA, Lang B, Oddis CV, van Royen A, Vencovsky J, Werth VP, Machado PM. Collaborative research in myositis-related disorders: MIHRA, a global shared community model. Clin Exp Rheumatol. 2024 Feb;42(2):207-212. doi: 10.55563/clinexprheumatol/hc1lsf. Epub 2024 Mar 4. PMID 38436382
- [Background] Lanis A, Alexanderson H, Ardalan K, Edison S, Graham CD, de Groot I, Gupta L, Kim S, Knight AM, Kobert L, Livermore P, Lood C, Pilkington C, Regardt M, Rubinstein TB, Shenoi S, Turnier L, Voet NBM, Wahezi DM, Saketkoo LA. Mental health in paediatric and adult myositis-related diseases: current state of research, interventions, and future steps from the MIHRA Psychological Impact Scientific Working Group. Clin Exp Rheumatol. 2024 Feb;42(2):413-424. doi: 10.55563/clinexprheumatol/cngdfn. Epub 2024 Mar 14. PMID 38488093
- [Background] Saketkoo LA, Valenzuela A, Kim S, McCann LJ, Lood C, Wahezi DM, Werth VP, Yi B, Alexanderson H, Maillard S, Pilkington C, Fligelstone K, Limbach B, Orandi AB, Regardt M, Russell AM, Davuluri S, deGroot I, Ernste F, Paik JJ, von Muhlen CA, Dimachkie MM, Machado PM, Naddaf E, Shafranski BM, Gupta L, Zulian F, Chung L; International Myositis Assessment and Clinical Studies Group and The Myositis International Research and Health Collaborative Alliance (IMACS/MIHRA) Calcinosis Scientific Interest Group. Moving forward together: collaborative landscapes of research in idiopathic inflammatory myopathies and calcinosis. Rheumatology (Oxford). 2024 May 2;63(5):1189-1191. doi: 10.1093/rheumatology/kead331. No abstract available. PMID 37449887
- See also: How to Participate through the MIHRA Patient Contact Registry — https://mihrafoundation.org/mihra-programs/mihra-patient-contact-registry/